CLINICAL TRIAL: NCT03187600
Title: Single Blinded Randomized Controlled Trial Comparing Muscular Pharyngeal Flap to Mucosal/Submucosal Pharyngeal Flap Surgical Technique for the Treatment of Velopharyngeal Dysfunction
Brief Title: Submucosa/Mucosal Pharyngeal Flap Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Murad Husein, aediatric Otolaryngologist Associate Professor and Undergraduate Director, Department of Otolaryngology-Head and Neck Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109037
Record Dates: First submitted 2017-06-11; First posted 2017-06-15 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Velopharyngeal Insufficiency
MeSH Terms: conditions — Velopharyngeal Insufficiency | interventions — Endomet

STUDY DESIGN:
Intervention Model Description: 1 group will receive a pharyngeal flap procedure comprised of pharyngeal muscle while the other group will receive of a procedure with only mucosa/submucosa.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be told what procedure they have received until after completion int he study. Speech language pathologists performing assessments will not be made aware of what procedure the patients have received. Nasovideo endoscopy will be reviewed in a blinded fashion without knowledge of what procedure the patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Procedure: a superiorly based pharyngeal flap surgery as per Hogan and Cable and Canady. It is performed trans-orally under general anesthetic. The soft palate is divided midline to visualize the posterior pharyngeal wall. A small flap is dissected via longitudinal incisions with a superior pedicle from the posterior pharyngeal wall at the level of the velum. The flap is then brought anteriorly, the inferior portion is lined with mucosa from the nasal portion of the soft palate and sutured in-place to create an incomplete pharyngeal obstruction that acts as a dynamic valve. Nasal stents are placed in each lateral port to prevent airway compromise and maintain flap integrity. Stents are removed two days post operatively and the patient is discharged after removal of stents and deemed to have a stable airway. Dissection will be carried out to the level of the prevertebral fascia and be comprised of mucosa and pharyngeal muscle.
  Interventions: Procedure: Standard of Care Pharyngeal Flap
- Experimental Group (Experimental): Procedure: a modified superiorly based pharyngeal flap surgery as per Hogan and Cable and Canady. It is performed trans-orally under general anesthetic. The soft palate is divided midline to visualize the posterior pharyngeal wall. A small flap is dissected via longitudinal incisions with a superior pedicle from the posterior pharyngeal wall at the level of the velum. The flap is then brought anteriorly, the inferior portion is lined with mucosa from the nasal portion of the soft palate and sutured in-place to create an incomplete pharyngeal obstruction that acts as a dynamic valve. Nasal stents are placed in each lateral port to prevent airway compromise and maintain flap integrity. Stents are removed two days post operatively and the patient is discharged after removal of stents and deemed to have a stable airway. Dissection will be carried out only to the level of the superior constrictor muscle and comprised of mucosua/submucosa
  Interventions: Procedure: Mucosa/submucosa Pharyngeal Flap

INTERVENTIONS:
Procedure: Mucosa/submucosa Pharyngeal Flap — Included in study arm description
  Arms: Experimental Group
Procedure: Standard of Care Pharyngeal Flap — Included in study arm description
  Arms: Standard of Care

SUMMARY:
The investigators want to compare two different surgical techniques for the treatment of a condition called velopharyngeal dysfunction (VPD). VPD is a condition in which the nasal part of the airway does not close properly during speaking and feeding. The current standard surgical management involves taking a pharyngeal flap from the back of the throat comprised of muscle and overlying mucosal tissue to create a functioning valve. The proposed technique would use only the mucosal/submucosal layer of the pharynx for the flap. This technique has been shown to be effective in animal models and it is hoped that it will lead to faster healing, lower complications and improved functional outcome for patients.

DETAILED DESCRIPTION:
Velopharyngeal dysfunction (VPD) results from failure of the airway to close and separate the oropharynx and nasopharynx during speech, eating and drinking as a result of insufficiency of the velum (soft palate) (1). VPD leads to a number of symptoms including difficulty with articulation, nasal regurgitation and excess nasal air emissions. VPD can often be treated through speech language therapy alone, however when refractory to this treatment surgical correction of problematic anatomy is indicated (2). The current surgery of choice at this center is a pedicled, posterior wall pharyngeal flap. During this procedure a small flap comprised of mucosa, submucosa and superior pharyngeal constrictor muscle is pedicled via surgical dissection and attached anteriorly to the inadequate soft palate. This creates an incomplete midline obstruction at the level of the velum allowing for a dynamic valve which can be closed through the medial constriction of the pharyngeal muscles during speech and eating/drinking. While this surgery has a high success rate there can be a high degree of post operative pain and sub-optimal lateral wall motion (2). It is hypothesized that the suboptimal lateral wall motion post-operatively is due to intentional segmentation of the superior constrictor muscle during the operation. Due to the necessary de-innervation of the pedicled pharyngeal flap there is evidence that the muscle atrophies and the bulk it initially adds to the flap is lost over time. Despite this, patients typically have good long-term outcomes with a pharyngeal flap (3,4). For these reasons it has been postulated that a successful surgery could be carried out using a pharyngeal flap comprised only of mucosa and submucosa, sparing the superior constrictor muscle. By sparing the superior constrictor muscle the investigators hope to achieve a decrease in post operative pain, complications and improved lateral wall motion while maintaining the effectiveness of the flap and symptomatic improvement. This novel surgical approach to treating VPD was shown to be effective and safe in animal trial (2). The major concern of the mucosal/submucosal flap procedure was that the flap would atrophy and fail without the inclusion of the muscular portion. However, results of the animal study comparing the standard pharyngeal flap to the experimental flap, indicated that at 12 weeks post-operation, bulk loss in the muscosa/submucosa group was not significantly greater than bulk loss in the muscular flap group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with velopharyngeal dysfunction undergoing pharyngeal flap surgery for correction.

Exclusion Criteria:

* Patients suffering VPD secondary to a syndrome. Patients undergoing a revision pharyngeal flap surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-06-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in Hypernasality | 3-4 months post-operatively
  The primary outcome of the study will be improvement of hypernasality assessed by the ACPA perceptual assessment

SECONDARY OUTCOMES:
ACPA Perceptual Assessment | 3-4 months post-operatively
  The remainder of the ACPA perceptual assessment (hyponasality, audible nasal emission, articulation proficiency, overall intelligibility, and compensatory articulation),
post-operative pain | 0-2 months post-operatively
  Post-op pain will be tracked using a validated pain scale as well as medication log.
complications associated with the procedure | 0-1 month post-operatively
  subjectively assessed

CONTACTS AND LOCATIONS:
Overall Officials: Murad Husein, MD, FRCSC, Principal Investigator — Lawson Heath Research Institute
Locations (1):
- Childrens Hospital London Health Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No